CLINICAL TRIAL: NCT03516461
Title: Efficacy and Safety of Fecal Microbiota Transplantation in Radiation Enteritis
Brief Title: Fecal Microbiota Transplantation for Radiation Enteritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Microbiota Medicine, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-RE-201702
Record Dates: First submitted 2018-01-07; First posted 2018-05-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Radiation Enteritis
Keywords: Gut Microbiota; Radiation Enteritis; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiota Transplantation (FMT) (Experimental): Patients receive a course of FMT during hospitalization
  Interventions: Procedure: Fecal Microbiota Transplantation (FMT)
- Basic treatment (No Intervention): Patient receives basic therapy for RE during hospitalization

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation (FMT) — Fecal microbiota transplantation for patients via nasointestinal tube or gastroscopy or colonic TET tube
  Other Names: FMT
  Arms: Fecal Microbiota Transplantation (FMT)

SUMMARY:
Radiation enteritis is one of the most feared complications after abdominal or pelvic radiation therapy.The gut microbiota is considered to constitute a "microbial organ" which has pivotal roles in the intestinal diseases and body metabolism. Evidence from animal studies demonstrated the link between intestinal bacteria and radiation enteritis. This clinical trial aims to evaluate the efficacy and safety of fecal microbiota transplantation (FMT) for radiation enteritis.

DETAILED DESCRIPTION:
The present clinical trial aims to re-establish a gut functionality state of intestinal microbiota through fecal microbiota transplantation (FMT) for radiation enteritis (RE). FMT is the whole profile of fecal microbiota transplantation. At enrollment, "Shared Decision Making" intervention was applied to support patient involvement in making health decisions. Patients have opportunity to choose fecal microbiota transplantation (FMT). Patients will receive follow-up for at least 12 weeks. Blood test, endoscopy and questionnaire will be used to access participants at study start and at study completion. Fecal microbiota compositions, blood and urinary metabolic profiles of patients will be analyzed to assess associated microbial changes.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old;
2. Radiation enteritis diagnosed by colonoscopy after finishing radiotherapy.

Exclusion Criteria:

1. Patients who were pregnant or nursing;
2. Patients who were unable or unwilling to undergo a gastroscopy;
3. Patients who had gastrointestinal infection;
4. Patients with cardiopulmonary failure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 12 weeks
  The clinical response rate at 8 weeks after fmt treatment

SECONDARY OUTCOMES:
Scores of gastrointestinal symptoms | 4, 8, 12 weeks
  Gastrointestinal symptoms will be evaluated according to NCI-CTC 5.0
Change of toxicity grade | 4, 8, 12 weeks
  The change of toxicity grade according to the RTOG/EORTC toxicity scale at 4, 8, 12 weeks after FMT

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD; PHD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cui M, Xiao H, Li Y, Zhou L, Zhao S, Luo D, Zheng Q, Dong J, Zhao Y, Zhang X, Zhang J, Lu L, Wang H, Fan S. Faecal microbiota transplantation protects against radiation-induced toxicity. EMBO Mol Med. 2017 Apr;9(4):448-461. doi: 10.15252/emmm.201606932. PMID 28242755
- [Background] Borody TJ, Khoruts A. Fecal microbiota transplantation and emerging applications. Nat Rev Gastroenterol Hepatol. 2011 Dec 20;9(2):88-96. doi: 10.1038/nrgastro.2011.244. PMID 22183182
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] Ferreira MR, Muls A, Dearnaley DP, Andreyev HJ. Microbiota and radiation-induced bowel toxicity: lessons from inflammatory bowel disease for the radiation oncologist. Lancet Oncol. 2014 Mar;15(3):e139-47. doi: 10.1016/S1470-2045(13)70504-7. PMID 24599929
- [Background] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757
- [Background] Manichanh C, Varela E, Martinez C, Antolin M, Llopis M, Dore J, Giralt J, Guarner F, Malagelada JR. The gut microbiota predispose to the pathophysiology of acute postradiotherapy diarrhea. Am J Gastroenterol. 2008 Jul;103(7):1754-61. doi: 10.1111/j.1572-0241.2008.01868.x. Epub 2008 Jun 28. PMID 18564125
- [Background] Wang A, Ling Z, Yang Z, Kiela PR, Wang T, Wang C, Cao L, Geng F, Shen M, Ran X, Su Y, Cheng T, Wang J. Gut microbial dysbiosis may predict diarrhea and fatigue in patients undergoing pelvic cancer radiotherapy: a pilot study. PLoS One. 2015 May 8;10(5):e0126312. doi: 10.1371/journal.pone.0126312. eCollection 2015. PMID 25955845
- [Background] Kim YS, Kim J, Park SJ. High-throughput 16S rRNA gene sequencing reveals alterations of mouse intestinal microbiota after radiotherapy. Anaerobe. 2015 Jun;33:1-7. doi: 10.1016/j.anaerobe.2015.01.004. Epub 2015 Jan 16. PMID 25600706
- [Background] Delia P, Sansotta G, Donato V, Messina G, Frosina P, Pergolizzi S, De Renzis C, Famularo G. Prevention of radiation-induced diarrhea with the use of VSL#3, a new high-potency probiotic preparation. Am J Gastroenterol. 2002 Aug;97(8):2150-2. doi: 10.1111/j.1572-0241.2002.05946.x. No abstract available. PMID 12190202
- [Background] Demers M, Dagnault A, Desjardins J. A randomized double-blind controlled trial: impact of probiotics on diarrhea in patients treated with pelvic radiation. Clin Nutr. 2014 Oct;33(5):761-7. doi: 10.1016/j.clnu.2013.10.015. Epub 2013 Oct 24. PMID 24200199
- [Background] Nascimento M, Aguilar-Nascimento JE, Caporossi C, Castro-Barcellos HM, Motta RT. Efficacy of synbiotics to reduce acute radiation proctitis symptoms and improve quality of life: a randomized, double-blind, placebo-controlled pilot trial. Int J Radiat Oncol Biol Phys. 2014 Oct 1;90(2):289-95. doi: 10.1016/j.ijrobp.2014.05.049. PMID 25304789
- [Derived] Ding X, Li Q, Li P, Chen X, Xiang L, Bi L, Zhu J, Huang X, Cui B, Zhang F. Fecal microbiota transplantation: A promising treatment for radiation enteritis? Radiother Oncol. 2020 Feb;143:12-18. doi: 10.1016/j.radonc.2020.01.011. Epub 2020 Feb 7. PMID 32044171